CLINICAL TRIAL: NCT05017051
Title: Study for the Quantification in Ecological Conditions of Sensorimotor and Dysexecutive Disorders in Cerebral Palsy Patients
Acronym: SDS2
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2018PPRC34; 2021-A00087-34 (Other: IDRCB)
Record Dates: First submitted 2021-08-19; First posted 2021-08-23 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Dysexecutive Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysexecutive patients: Patients with dysexecutive syndrome
  Interventions: Behavioral: Chocolate cake; Behavioral: Lego model; Device: Measurement of sensorimotor abilities; Other: Measurement of facial expression of emotions
- Healthy subjects: Healthy subjects to be used as control group
  Interventions: Behavioral: Chocolate cake; Behavioral: Lego model; Device: Measurement of sensorimotor abilities; Other: Measurement of facial expression of emotions

INTERVENTIONS:
Behavioral: Chocolate cake — The participants will have to make a chocolate cake following an imposed recipe at 4 visits (initially (M0), after 12 months (M12), after 24 months (M24) and after 36 months (M36)).
Behavioral: Lego model — The participants will have to build a Lego model at 4 visits (M0, M12, M24 and M36).
Device: Measurement of sensorimotor abilities — The measurement of sensorimotor abilities is based on a multi-sensor device called Smart Flat specifically designed for this study at 4 visits (M0, M12, M24 and M36).
Other: Measurement of facial expression of emotions — Participants will have to evoke an emotionally charged autobiographical story by modulating facial expressions through a mirror at 4 visits (M0, M12, M24 and M36).

SUMMARY:
Executive functions are defined as the mental functions necessary for an individual to adapt to a complex or new environment that requires freedom from automatic and routine behavior. Deficits in executive functions are described under the term "dysexecutive syndrome", and call into question the quality of social and professional life as well as the autonomy of patients.

The usual methods of identifying dysexecutive syndrome are based essentially on batteries of neuropsychological tests known as "paper and pencil". However, these tests may lack sensitivity, in that they assess the patient in a very structured setting, very different from real life conditions, which are full of distractions and choices to be made.

Evaluations on real tasks are more rarely used but have the advantage of observing the difficulties encountered by a patient in everyday life.

Two tests of this type have been set up in the Neurology Department of the Hôpital d'Instruction des Armées Percy, and are integrated into the routine care of patients with a dysexecutive syndrome.

For this purpose, a room in the department has been set up as a studio in order to reproduce as much as possible an everyday life environment, in which executive functions, fine motor skills, neurovegetative functions, emotional state, posture, locomotor skills and visual information capture can be measured ecologically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a dysexecutive syndrome OR healthy subjects
* Over 18 years-old

Exclusion Criteria:

* Patients

  * Psychiatric pathology (except for Post-Traumatic Stress Disorder)
  * Pregnant or breastfeeding woman
* Healthy subjects

  * Neurologic or psychiatric pathology
  * Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of 2 groups:
  * a group of patients with dysexecutive syndrome
  * a group of healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 442 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Lowest number of errors on the executive tasks over the 4 visits | Until the end of the study (3 years)
  An error is defined as: an omission, an addition, a substitution, an estimation error, a question or a commentary The number of errors will be calculated for each task at each visit. The lowest number will be retained to compare the 2 groups.

SECONDARY OUTCOMES:
Lowest number of errors on the Lego model task over the 4 visits | Until the end of the study (3 years)
  An error is defined as: an omission, an addition, a substitution, an estimation error, a question or a commentary
  The number of errors will be calculated for the Lego model task at each visit. The lowest number will be retained to compare the 2 groups.
Lowest number of errors on the chocolate cake task over the 4 visits | Until the end of the study (3 years)
  An error is defined as: an omission, an addition, a substitution, an estimation error, a question or a commentary
  The number of errors will be calculated for the chocolate cake task at each visit.
  The lowest number will be retained to compare the 2 groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Percy, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided